CLINICAL TRIAL: NCT02097615
Title: Clinical Trial of the Effectiveness of Chlorhexidine Gluconate 0.125 % Compared With Sterile Deionized Water in the Closure of Diabetic Foot Ulcer Syndrome.
Brief Title: Diabetic Foot Ulcer. Effectiveness of Chlorhexidine Gluconate 0.125 % Compared With Sterile Deionized Water
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Alejandro E. Macias, Physician, Universidad de Guanajuato
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GTSSA02101-298
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2014-12

CONDITIONS: Soft Tissue Infections
Keywords: soft; tissue; infections
MeSH Terms: conditions — Soft Tissue Infections; Infections | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chlorhexidine gluconate (Experimental): application every 24 hours, six weeks
  Interventions: Procedure: chlorhexidine gluconate
- Other: deionized water (Other): application every 24 hours, six weeks
  Interventions: Other: deionized water

INTERVENTIONS:
Procedure: chlorhexidine gluconate — chlorhexidine gluconate spray of 0.125% . Application in the area of the ulcer every 24 hours for six weeks
  Arms: chlorhexidine gluconate
Other: deionized water — application every 24 hours six weeks
  Arms: Other: deionized water

SUMMARY:
At present research has generated controversy regarding the utility of antiseptics in wound management for diabetic foot ulcers syndrome. However, these studies have been done in tissues and animal models. This study involves the best presently antiseptic for residual effect and low toxicity in an approach to eliminate microorganisms promoters formation of biofilm, contributing to the treatment for accelerated closure the diabetic foot ulcers syndrome .

So it is necessary to determine if irrigation ulcer diabetic foot syndrome with chlorhexidine 0.125 % aqueous solution determines the decrease of the surface to a greater extent than the standard treatment using irrigation with sterile deionized water .

DETAILED DESCRIPTION:
The present study be made performed at the Hospital General Leon.

Population:

People with Diabetes Mellitus state of Guanajuato.

Universe:

People with diabetes mellitus and diabetic foot syndrome Guanajuato state . sample: Will be evaluated in patients with diabetes mellitus presenting loss of continuity of the skin of the lower limbs and coming to the clinic wound´s of the León General Hospital . This clinic provides services to patients in the state of Guanajuato with diabetic foot syndrome, including them within a multidisciplinary management program .

Calculation of Sample :

72 patients; more eight for lost estimates, 40 patients for each group are required to have a 80 % chance of detecting , with a significance level of 5%, an increase in the primary outcome measure of 5% in the control group and 6 % in group experimental .

Alpha: 5 % Power : 80 %

Inclusion Criteria:

Indistinct gender Patients over 18 years with Diabetes Mellitus and submit ulcer from diabetic foot syndrome not involving tendon , capsule or bone.

With proper state of vascular perfusion.

Exclusion Criteria :

Ulcers in patients with interdigital or difficult to measure the affected surface areas.

Patients not be located at follow-up or wish to stop participating in the study.

Methodology:

Will be invited to participate in the study patients with diabetes mellitus consecutive presented with ulcers plantar to IA or IB grade classification system ulcers , University of Texas, in the area of Clinical wound´s of the Hospital General Leon between Abril and November 2014.

After explaining the study information and check which is understandable , they provide the sheet to be signed informed consent.

Subsequently selected patients will be given a vascular ultrasound to measure the ankle brachial index and determine the absence of vascular compromise.

They carry out their medical history with emphasis on analyzing clinical data , including the characteristics of the ulcer (type of exudate , measured surface area affected , type of tissue involved in the ulcer to its depth ) and biochemical parameters .

Be weighed and measured at the first visit and not having biochemical data are requested to collect this information in subsequent follow-up visit .

They were then treated with the principles of the standard treatment, under the following criteria :

* Remove the ulcer exudate by spraying one of the two ingredients making mechanical drive for 5 minutes, or until completely negative to the visual evidence of exudate.
* Completely remove hyperkeratosis and devitalized tissue from the periphery of the ulcer with cutting material dissection with sterile dressing and drag , until visually eliminate the exudate.
* The treated area is dry and sore
* Two photographs at a distance of 20 cm perpendicular to the ulcer will be taken, covering a 1 square centimeter reference for measuring the area affected by diabetic foot ulcer syndrome.
* The solution so blinded to the ulcer and covered with sterile dressing will be applied for 24 hours .
* The patient will be instructed to continue treatment every 24 hours as follows :
* Sterile dressing will be removed and continuously irrigate for 5 seconds with the ingredient that was assigned .
* Undiscovered for 24 hours , until the next day irrigation dressing area will be placed . Also need to avoid contact with any surface over the affected area until the next assessment .
* Perform the same strategy for 24 hours , and on day 7 will go to the wound clinic to clinical evaluation.
* Every 7 days until complete 6 views, clinical evaluation are performed, irrigation with the selected ingredient and it will take 2 pictures at a distance of 20 cm perpendicular to the boil again , covering a reference of 1 square centimeter to measure the area affected by the diabetic foot ulcer syndrome.
* Every 7 days of initiation of therapy in the clinic consultation wounds measured and circulation and comment the following:
* Ulcer area in square millimeters .
* Coloring of the ulcer .
* Type of exudate ; turbid serous .
* Type of tissue involved in the ulcer to its depth. If any patients have increased intensity of the signs and symptoms of diabetic foot syndrome, classified as a major step on the scale of ulcers Classification System of the University of Texas, perform analysis and comprehensive treatment will be redefined according to the suggestions of ulcer classification system of the University of Texas.

Material cleaning the ulcer :

Ingredient 1: Preparation of spray application of chlorhexidine gluconate 0.125% .

Ingredient 2: Preparation of spray application of sterile deionized water .

Method of application of ingredients as described previously .

Method of randomization : is effected by assigning random numbers balanced computer, the code will be assigned to each of the ingredients which have identical presentations , they will balance to the sample size . The code will not be known by the patient, observer and analyst. Only be known by one of the advisors.

Statistical methods :

The description of the data, in the case of non-numerical variables will be performed by reporting proportions and confidence interval of 95 % (95 %) in the case of numerical variables, the description will be made based on averages and standard deviation or medians and Q1- Q3 range , depending on the result of the Kolmogorov-Smirnov test to evaluate the Gaussian distribution of the data.

Comparison of numerical variables were not performed by Chi square test . Comparison of the rates of reduction in the size of ulcers of diabetic foot syndrome for both treatments will be based on the t test for independent samples or by Kruskal- Wallis test , depending on data distribution .

In all cases be considered as the significance level alpha value <0.05 .

ELIGIBILITY:
Inclusion Criteria:

* Indistinct gender
* Patients over 18 years with Diabetes Mellitus and
* Submit ulcer from diabetic foot syndrome not involving tendon , capsule or bone.
* With proper state of vascular perfusion.

Exclusion Criteria:

* Ulcers in patients with interdigital or difficult to measure the affected surface areas.
* Patients not be located at follow-up or wish to stop participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Unlike the ultimate determinations for the initial surface of the ulcer obtained in square millimeters. | 15 days
  Total ulcer area shall be measured by drawing software AUTOCAD LT 2014 , which defines the edges of the ulcer surface area in each of the two photographs , to take an average of the measure and get a value to be analyzed, that value is checked against the reference area of 1 square centimeter to increase measurement accuracy .

CONTACTS AND LOCATIONS:
Overall Officials: Hugo A Manriquez Perez, Physician, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Hospital General Leon, León, Guanajuato, Mexico